CLINICAL TRIAL: NCT00670475
Title: Comparative Study of Olive Oil With Piroxicam Gel in Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ardabil University of Medical Sciences (Other)
Responsible Party: Shahab Bohlooli, pharmacology dept, faculty of medicine, ArdabilUMS
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1/86010
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2010-04-29 (Estimated); Status verified 2010-04

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis; Knee; virgin olive oil; piroxicam; Topical
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Piroxicam; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- P (Pircoxicam Group) (Active Comparator): in this arm 100 patients with osteoarthritis of knee will receive piroxicam gel in blinded 60 grams tubes,they will be instructed to use 1 gram of piroxicam gel (with inserted dispensing device) three times in a day on the affected knee.
  Interventions: Drug: Piroxicam
- O (olive oil group) (Experimental): in this arm 100 patients with osteoarthritis of knee will receive virgin olive oil in blinded 60 grams tubes,they will be instructed to use 1 gram of olive oil (with inserted dispensing device) three times in a day on the affected knee.
  Interventions: Dietary Supplement: Olive Oil

INTERVENTIONS:
Drug: Piroxicam — In this interventional arm gel of piroxicam (manufactured by Iran najo co,Iran), repackaged in a 60 g anonymous tubes will be administered to the patients.
  Other Names: Piroxicam topical gel
  Arms: P (Pircoxicam Group)
Dietary Supplement: Olive Oil — virgin olive oil prepared directly from olive fruit from "olive gardens of north of iran, Gilan province" will packaged in a 60 g anonymous tubes.
  Other Names: Topical virigin olive oil
  Arms: O (olive oil group)

SUMMARY:
this is a randomized double blinded trial which is conducted to measure the efficacy of topical virgin olive oil on osteoarthritis of knee that will be done in contrast to standard piroxicam gel.

DETAILED DESCRIPTION:
application of herbal product has old history in therapy of human diseases. olive oil is one of the important diet in Iran which its efficacy in reducing of rheumatic pains was pointed out by Avicenna in 10th century. Nevertheless, its efficacy is not confirmed by scientific study.

in this double blinded study, 200 patients with diagnosed osteoarthritis of knee will be recruited that will randomly be assigned in piroxicam or olive oil group. the piroxicam gel or olive oil will be repackaged in anonymous tubes, which only recognizable via codes. the patients or visiting clinicians will be unaware of content of tubes. the final assessor will be blind to groups and interventions.

the efficacy of therapies will be evaluated by means of WOMAC and PGs standard questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* men and non-pregnant women, age 40-85 years with primary OA of at least one knee, and a flare of pain after withdrawal of prior therapy with either an oral NSAID or acetaminophen (used at least 3 days per week during the previous month).

Exclusion Criteria:

* secondary arthritis related to systemic inflammatory arthritis (including rheumatoid arthritis, psoriatic arthritis, post-infectious arthritis and metabolic arthritis, traumatic arthritis or surgical joint replacement); corticosteroid use:

  * oral corticosteroid within the previous 14 days, or
  * intramuscular corticosteroid within 30 days, or
  * intraarticular corticosteroid into the study knee within 90 days,
  * intra-articular corticosteroid into any other joint within 30 days, or
  * topical corticosteroid at the site of application within 14 days;
* ongoing use of prohibited medication including NSAID, other oral analgesic, muscle relaxant, or low-dose antidepressant for any chronic pain management; - ongoing use of glucosamine or chondroitin (unless used continuously for 90 days prior to study entry);
* sensitivity to diclofenac, acetylsalicylic acid (ASA) or any other NSAID, acetaminophen, dimethyl sulphoxide, propylene glycol, glycerine or ethanol; clinically-active renal, hepatic or peptic ulcer disease;
* history of alcohol or drug abuse;
* lactation;
* concomitant skin disease at the application site;
* current application for disability benefits on the basis of knee osteoarthritis; fibromyalgia; other painful or disabling condition affecting the knee;

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures is defined as the change from baseline to final assessment of the study knee in the 3 core continuous variables pain and physical function, assessing using the WOMAC subscales, and patient global assessment (PGA). | the outcome is assessed at week 1
The primary outcome measures is defined as the change from baseline to final assessment of the study knee in the 3 core continuous variables pain and physical function, assessing using the WOMAC subscales, and patient global assessment (PGA). | the outcome is assessed at week 2
The primary outcome measures is defined as the change from baseline to final assessment of the study knee in the 3 core continuous variables pain and physical function, assessing using the WOMAC subscales, and patient global assessment (PGA). | the outcome is assessed at week 3
The primary outcome measures is defined as the change from baseline to final assessment of the study knee in the 3 core continuous variables pain and physical function, assessing using the WOMAC subscales, and patient global assessment (PGA). | the outcome is assessed at week 4

SECONDARY OUTCOMES:
the secondary measure will be changes in stiffness | the outcome is assessed at week 1
the secondary measure will be changes in stiffness | the outcome is assessed at week 2
the secondary measure will be changes in stiffness | the outcome is assessed at week 3
the secondary measure will be changes in stiffness | the outcome is assessed at week 4

CONTACTS AND LOCATIONS:
Overall Officials: shahab bohlooli, PhD, Principal Investigator — Pharmacology Dept, Faculty of Medicine, ArdabilUMS; Marina Jastan, MD, Principal Investigator — rheomatology clinic, faculty of medicine, ArdabilUMS
Locations (1):
- ArdabiUMS clinic of rheumatology, Ardabil, Ardabil Province, Iran